CLINICAL TRIAL: NCT01300117
Title: Influence of Extracorporeal Circulation During Cardiac Surgery on the Development of Postoperative TTP
Brief Title: Influence of Extracorporeal Circulation During Cardiac Surgery on the Development of Postoperative Thrombotic Thrombocytopenic Purpura (TTP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Dr. med. W. Miesbach, Hämophilie Zentrum, JWG University Hospital
Other Study IDs: TTP-KC
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; adamts13; TTP; extracorporeal circulation; Heart-Lung Machine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with extracorporeal circulation: Patients undergoing cardiac surgery with the use of an extracorporeal circulation
- without extracorporeal circulation: Patients undergoing cardiac surgery without the use of extracorporeal circulation (OPCAB)

SUMMARY:
The purpose of this study is to determine whether extracorporeal circulation during cardiac surgery has an influence on ADAMTS13-Activity.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgery with or without (OPCAB) the use of extracorporeal circulation
* patient agrees

Exclusion Criteria:

* no agreement
* known TTP in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery at the University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
Change in ADAMTS13-Activity over time | during surgery (at 1and 2 hours after beginning) and within the first 6 days after surgery

SECONDARY OUTCOMES:
Change in ADAMTS13-Antibody over time | during surgery (at 1and 2 hours after beginning) and within the first 6 days after surgery
Change in Platelet count over time | during surgery (at 1and 2 hours after beginning) and within the first 6 days after surgery
time duration of extracorporeal circulation during surgery | during surgery
Amount of intraoperative given fluid replacement | during surgery
Amount of given blood products (red blood cells) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Hesse, Germany